CLINICAL TRIAL: NCT03105466
Title: Prospective Study of Deep Anterior Lamellar Keratoplasty Using Acellular Porcine Cornea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jin Yuan, Professor, Zhongshan Ophthalmic Center, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016021
Record Dates: First submitted 2016-08-31; First posted 2017-04-10 (Actual); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Corneal Transplantation
Keywords: Corneal Transplantation; Xenotransplantation; Bioegineered cornea

ARMS (1):
- Acellular porcine cornea group (Experimental): Participants with corneal diseases not involving the endothelial layer undergo deep anterior lamellar keratoplasty using acellular porcine cornea
  Interventions: Procedure: Deep anterior lamellar keratoplasty; Device: Acellular Porcine Cornea; Drug: Tacrolimus eye drops; Drug: Tobradex eyedrops

INTERVENTIONS:
Procedure: Deep anterior lamellar keratoplasty — Deep anterior lamellar keratoplasty using acellular porcine cornea; 0.05%Tacrolimus eye drops, four times a day for at least one year; 0.3% Tobradex eyedrops, four times-one times a day for one year.
Device: Acellular Porcine Cornea
Drug: Tacrolimus eye drops
Drug: Tobradex eyedrops

SUMMARY:
The performance of keratoplasty is hampered by the limited availability of donor cornea in many countries, especially in Asia. For this reason, attempts have been made to fabricate artificial substitutes for natural human cornea. So far, all polymeric biomaterials, such as collagen configurations and plastic compression, could mimic the functional optically transparent but failed to replicate the complicate three-dimension microstructure of natural cornea. Therefore, despite some favorable results yielded by polymeric biomaterials, they cannot be suited for long-term use. To overcome these disadvantages, in recent years, porcine cornea appeared specifically attractive for xenotransplantation, because of its accessibility and similarities to natural human cornea. However, xenotransplantation using fresh porcine cornea can occurs hyperacute immune rejection, resulting in graft failure. Such transplant rejection can be substantially lessened by using acellular porcine cornea (APC), which preserves the constructure of natural cornea, whilst having well biocompatibility and low antigenicity. These properties feature APC particularly suitable for high-risk keratoplasty, such as corneal grafting in infectious keratitis.

Use of APC in LK has been shown promise in many preclinical animal studies and initially in human clinic trail. However, to optimize APC biological and biomechanical properties, the strategies for its preparation has evolved extensively over recent years, like various decellularization approaches (e.g. detergents, enzymes, human sera, hypertonic solutions and et al) and additional procedures (e.g. collagen re-crosslinking and repeated frozen-dry). Therefore, in the current study, the investigators analyzed the early surgical outcomes of deep anterior lamellar keratoplasty (DALK) using the APC that was very recently approved by the National Institutes for Food and Drug Control (NIFDC) of China for clinic practice, for management of infective keratitis, including fungal, viral and acanthamoeba keratitis. Here major concern of this study was to clarify the behavior of APC after implantation in participants.

ELIGIBILITY:
Inclusion Criteria:

corneal diseases not involving the endothelial layer

Exclusion Criteria:

* corneal diseases involving the endothelial layer
* allergic to pig tissue
* do not accept xenotransplantation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-02; Primary Completion 2020-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
the changes of Best corrected visual acuity | Before surgery, 1-week, 1-month, 3-month, 6-month, 1-year, 2-year, 3-year, 4-year after surgery

SECONDARY OUTCOMES:
the changes of visual contrast sensitivity | Before surgery, 3-month, 6-month, 1-year, 2-year, 3-year, 4-year after surgery
the changes in the transparency of graft | 1-week, 1-month, 3-month, 6-month, 1-year, 2-year, 3-year, 4-year after surgery
  using Slit lamp microscopic evaluation
The changes in corneal thickness depth | 1-week, 1-month, 3-month, 6-month, 1-year, 2-year, 3-year, 4-year after surgery
  using anterior segmental OCT
The changes in corneal nerve regeneration | 1-month, 3-month, 6-month, 1-year, 2-year, 3-year, 4-year after surgery
  using Confocal microscopy
The changes of depression and anxiety status | Before surgery, 1-month, 3-month, 6-month, 1-year, 2-year, 3-year, 4-year after surgery
  Using Self-Rating Depression Scale (SDS) and Self-Rating Anxiaty Scale (SAS)

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-Sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Li S, Li M, Gu L, Peng L, Deng Y, Zhong J, Wang B, Wang Q, Xiao Y, Yuan J. Risk factors influencing survival of acellular porcine corneal stroma in infectious keratitis: a prospective clinical study. J Transl Med. 2019 Dec 30;17(1):434. doi: 10.1186/s12967-019-02192-z. PMID 31900186